CLINICAL TRIAL: NCT04969705
Title: Intrathecal Dexmedetomidine Versus Transversus Abdominus Plane Block (TAP) for Postoperative Analgesia After Cesarean Section.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Dina Mostafa Helmy, resident doctor, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-07-03
Record Dates: First submitted 2021-07-13; First posted 2021-07-21 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Pain Management in Adult Females in Child Bearing Period Aging From 20 to 45 Years Who Are Scheduled for Elective Cesarean Section
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (spinal Dexmedetomidine) (Active Comparator): . Spinal needles (22 G) will be introduced in sitting position after skin disinfection with povidine iodine, iliac crest will be palpated and thumb extended to meet the midline, feeling the space between L4 and L5. spinal needle penetrates through the dura matter, a pop will be felt and then after the needle puncture into the subarachnoid space and the appearance of clear cerebrospinal fluid, the intrathecal local anesthetic will be injected. All patients will be receiving 2 ml heavy bupivacaine 0.5% plus 5 µg dexmedetomidine to total volume of 2.5 ml.
  Interventions: Drug: Dexmedetomidine
- Group B (spinal with transversus abdominus plane block) (Active Comparator): Spinal needles (22 G) introduced in sitting position . patients receiving1.7 to 2.2 ml heavy bupivacaine 0.5%( according to weight and height ) + 1 ml normal saline = total volume of 2.5 ml then at surgery end under sonographic guide transducer placed in transverse plane above iliac crest.A 90 mm 22 G short beveled block needle inserted in-plane with transducer, in anterior-posterior direction. needle connected to syringe contains20 ml of bupivacaine 0.25%+10 µg dexmedetomidine to deposit local anesthetic deep into the fascial layer between internal oblique & transversus abdominis muscles on each side.
  Interventions: Drug: Dexmedetomidine
- Group C ( controlled group ) Spinal Anesthesia only : (Active Comparator): Patients will be anesthetized only with spinal anesthesia using Bupivacaine Hcl( 10 mg).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — 60 Patients will be randomly divided into three equal groups:
  Group A (n=20) : spinal anesthesia with Dexmedetomidine (5µg ) added to local anesthetic (bupivacaine Hcl ) (10 mg) given intrathecally .
  Group B (n=20) : spinal anesthesia using local anesthetic( bupivacaine Hcl) (20 mg) combined with TAP block using Dexmedetomidine (20µg ) after the cesarean section
  Group C (n=20) (controlled group ) : Spinal anesthesia using only local anesthetic (bupivacaine Hcl ) (10 mg) .

SUMMARY:
Spinal anesthesia is the most commonly used technique for lower abdominal surgeries as it is very economical and easy to administer. However, postoperative pain control is a major problem because spinal anesthesia using only local anesthetics is associated with relatively short duration of action, and thus early analgesic intervention is needed in the postoperative period The transversus abdominus plane (TAP) block is a regional analgesic technique which blocks T6-L1 nerve branches and has an evolving role in postoperative analgesia for lower abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status classes I and II
2. Scheduled for elective cesarean section
3. Aged between 20-45 years .

Exclusion Criteria:

1. patient refusal.
2. patient with significant cardiovascular disease , hepatic dysfunction , renal failure , chronic pulmonary disease .
3. neuromuscular disorder.
4. infection.
5. bleeding disorder.
6. Obesity ( BMI > 30 kg/m2 ) .
7. History of allergy or sensitivity to any of the study drugs in previous surgeries .

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Analgesic efficacy of both routes | 24 hours
  Demographic data (age, weight, and length), mean arterial blood pressure (MAP), and heart rate (HR) will be measured every 5 minutes intraoperatively and at 1, 2, 4, 6, 8,12,16,20 and 24 h postoperatively. Visual analog pain score (VAS) between 0 and 10 (0=no pain, 1-3=mild pain, 4-6=moderate pain, and 7-10=severe pain) will be recorded at 1, 2, 4, 6, 8,16,20 and 24 h postoperatively. First time of rescue analgesia: this is defined as the time from onset of sensory block till the time of first requirement of analgesia. The total amount of rescue analgesia consumption in the form of intravenous ketorolac→0.5 mg/kg if VAS greater than or equal to 4. Any undesirable postoperative side effects (as nausea, vomiting and pruritus) will be recorded and managed.

SECONDARY OUTCOMES:
1. Hemodynamic effect on the patient | 1 hour
  measuring BP , HR , oxygen saturation during operation every 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Betran AP, Merialdi M, Lauer JA, Bing-Shun W, Thomas J, Van Look P, Wagner M. Rates of caesarean section: analysis of global, regional and national estimates. Paediatr Perinat Epidemiol. 2007 Mar;21(2):98-113. doi: 10.1111/j.1365-3016.2007.00786.x. PMID 17302638
- [Background] Madadi P, Ross CJ, Hayden MR, Carleton BC, Gaedigk A, Leeder JS, Koren G. Pharmacogenetics of neonatal opioid toxicity following maternal use of codeine during breastfeeding: a case-control study. Clin Pharmacol Ther. 2009 Jan;85(1):31-5. doi: 10.1038/clpt.2008.157. Epub 2008 Aug 20. PMID 18719619
- [Background] Elia N, Culebras X, Mazza C, Schiffer E, Tramer MR. Clonidine as an adjuvant to intrathecal local anesthetics for surgery: systematic review of randomized trials. Reg Anesth Pain Med. 2008 Mar-Apr;33(2):159-67. doi: 10.1016/j.rapm.2007.10.008. PMID 18299097